CLINICAL TRIAL: NCT03802071
Title: A Phase I/II Study of Durvalumab in Combination With Standard Chemotherapy Doxorubicin for Advanced Soft Tissue Sarcoma
Brief Title: A Study of Durvalumab in Combination With Doxorubicin for Advanced Soft Tissue Sarcoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Hyo Song Kim, professor, Yonsei University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2018-0746
Record Dates: First submitted 2019-01-07; First posted 2019-01-14 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab+doxorubicin combination (Experimental)
  Interventions: Drug: Durvalumab+doxorubicin cobination

INTERVENTIONS:
Drug: Durvalumab+doxorubicin cobination — Durvalumab 1500mg IV Doxorubicin 75mg/m2 IV D1 Q3weeks (up to 8cycles)

SUMMARY:
The yearly incidence of soft-tissue sarcomas (STS) in the USA is roughly 11,280 cases, and metastatic STS have a median overall survival of about 12 months. Sarcomas of the soft tissue are a heterogeneous group of malignant tumors of mesenchymal origin that originate in connective tissue. Local control with wide surgical resection with or without adjuvant radiation has a success rate of close to 90%. However, approximately 40% to 50% of patients with a large (>5 cm), deep, high-grade soft-tissue sarcoma eventually develop distant metastases, primarily in the lung. Therefore, overall survival of metastatic STS remained still poor, less than 1 year. Therefore, current clinical trials with various targeted agents are ongoing add on the doxorubicin monotherapy.

Investigator planned to conduct the phase I/II trial of durvalumab in combination with standard chemotherapy, doxorubicin for metastatic/recurred sofe tissue sarcoma.

DETAILED DESCRIPTION:
The yearly incidence of soft-tissue sarcomas (STS) in the USA is roughly 11,280 cases, and metastatic STS have a median overall survival of about 12 months. Sarcomas of the soft tissue are a heterogeneous group of malignant tumors of mesenchymal origin that originate in connective tissue. Local control with wide surgical resection with or without adjuvant radiation has a success rate of close to 90%. However, approximately 40% to 50% of patients with a large (>5 cm), deep, high-grade soft-tissue sarcoma (STS) eventually develop distant metastases, primarily in the lung. Therefore, overall survival (OS) of metastatic STS remained still poor, less than 1 year. Therefore, current clinical trials with various targeted agents are ongoing add on the doxorubicin monotherapy.

Durvalumab (MEDI4736) is a human monoclonal antibody that inhibits binding of PD-L1. For this orphan tumor, STS, PD-L1 may be a promising strategy and favorable toxicity may warrant further combination. For this orphan tumor, STS, PD-L1 targeting may be a promising strategy and favorable toxicity may warrant further combination. Regarding anti-PD-L1 treatment in STS, in phase I trial with human monoclonal antibody to PD-L1, MPDL3280A, one heavily treated synovial sarcoma patients demonstrated partial responses. In recent phase II study of pembrolizumab, PD-1 inhibitor in advanced STS among the 40 STS cases (17.5%) had responses (1 complete response and 6 partial response). Based on the study, pembrolizumab monotherapy was approved for previously treated STS in Korea.

Therefore, various clinical trials are ongoing immune checkpoint inhibitor with PDGFR inhibitors [axitinib for renal cell carcinoma (RCC), pazopanib for RCC and STS, Sorafenib for RCC, and liver cancer, sunitinib for RCC, gastrointestinal stromal tumor, and pancreatic cancer].

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed STS(soft tissue sarcoma)
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
3. Measurable disease by Response Evaluation Criteria in Solid Tumors Version 1.1
4. Body weight >30kg
5. Adequate normal organ and marrow function as defined below:
6. Left ventricular ejection fraction (LVEF) ≥ 45%
7. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause.
8. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
9. Must have a life expectancy of at least 12 weeks
10. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations

Exclusion Criteria:

1. Histologically- or cytologically-confirmed Kaposi's sarcoma or GIST
2. Previous treatment with anthracyclines
3. Participation in another clinical study with an investigational product during the last 2 weeks
4. Receipt of the last dose of anticancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) 14 days prior to the first dose of study drug
5. Any previous treatment with a PD1 or PD-L1 inhibitor (including durvalumab) and/or PDGFR inhibitor
6. Mean QT interval corrected for heart rate (QTc) > 480 ms calculated from 3 electrocardiograms (ECGs) using Fridericia's Correction
7. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria
8. Any concurrent chemotherapy, biologic, or hormonal therapy for cancer treatment within 14 days prior to entering the study. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable
9. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 14 days of the first dose of study drug
10. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP(investigational product).
11. History of allogenic organ transplantation.
12. Active or prior documented autoimmune or inflammatory disorders
13. Uncontrolled intercurrent illness
14. Known active infection
15. History of another primary malignancy
16. History of leptomeningeal carcinomatosis who are neurologically unstable or have required active treatment
17. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP.
18. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose.
19. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2019-09-16 (Actual); Primary Completion 2022-08-10 (Estimated); Study Completion 2022-08-10 (Estimated)

PRIMARY OUTCOMES:
adverse event | 3 weeks
  to evaluate the safety and tolerability of durvalumab in combination with doxorubicin

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea